CLINICAL TRIAL: NCT05118789
Title: A Phase 1/2 Study of the Highly Selective ROS1 Inhibitor Zidesamtinib (NVL-520) in Patients With Advanced NSCLC and Other Solid Tumors (ARROS-1)
Brief Title: A Study of Zidesamtinib (NVL-520) in Patients With Advanced NSCLC and Other Solid Tumors Harboring ROS1 Rearrangement (ARROS-1)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nuvalent Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NVL-520-01
Record Dates: First submitted 2021-10-19; First posted 2021-11-12 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Solid Tumor; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1 dose escalation (Experimental): Zidesamtinib (NVL-520) oral daily dosing
  Interventions: Drug: Zidesamtinib (NVL-520)
- Cohort 2a (Experimental): ROS1+ NSCLC naïve to TKI therapy and up to 1 prior chemotherapy and/or immunotherapy
  Interventions: Drug: Zidesamtinib (NVL-520)
- Cohort 2b (Experimental): ROS1+ NSCLC treated with 1 prior ROS1 TKI and no prior chemotherapy or immunotherapy
  Interventions: Drug: Zidesamtinib (NVL-520)
- Cohort 2c (Experimental): ROS1+ NSCLC treated with 1 prior ROS1 TKI and 1 prior platinum-based chemotherapy with or without immunotherapy
  Interventions: Drug: Zidesamtinib (NVL-520)
- Cohort 2d (Experimental): ROS1+ NSCLC treated with ≥2 prior ROS1 TKIs and up to 1 prior chemotherapy and/or immunotherapy
  Interventions: Drug: Zidesamtinib (NVL-520)
- Cohort 2e (Experimental): ROS1+ solid tumor and progressed on any prior therapy
  Interventions: Drug: Zidesamtinib (NVL-520)

INTERVENTIONS:
Drug: Zidesamtinib (NVL-520) — Oral tablet of zidesamtinib (NVL-520)

SUMMARY:
Phase 1/2, dose escalation and expansion study designed to evaluate the safety and tolerability of zidesamtinib (NVL-520), determine the recommended phase 2 dose (RP2D), and evaluate the antitumor activity in patients with advanced ROS1-positive (ROS1+) NSCLC and other advanced ROS1-positive solid tumors.

Phase 1 will determine the RP2D and, if applicable, the maximum tolerated dose (MTD) of zidesamtinib in patients with advanced ROS1-positive solid tumors.

Phase 2 will determine the objective response rate (ORR) as assessed by Blinded Independent Central Review (BICR) of zidesamtinib at the RP2D. Secondary objectives will include the duration of response (DOR), time to response (TTR), progression-free survival (PFS), overall survival (OS), and clinical benefit rate (CBR) of zidesamtinib in patients with advanced ROS1-positive NSCLC and other solid tumors.

DETAILED DESCRIPTION:
In Phase 2, study patients will be enrolled into 5 distinct expansion cohorts:

* Cohort 2a: ROS1-positive NSCLC naïve to Tyrosine Kinase Inhibitor (TKI) therapy and up to 1 prior chemotherapy and/or immunotherapy.
* Cohort 2b: ROS1-positive NSCLC treated with 1 prior ROS1 TKI and no prior chemotherapy or immunotherapy.
* Cohort 2c: ROS1-positive NSCLC treated with 1 prior ROS1 TKI and 1 prior platinum-based chemotherapy with or without immunotherapy.
* Cohort 2d: ROS1-positive NSCLC treated with ≥2 prior ROS1 TKIs and up to 1 prior chemotherapy and/or immunotherapy.
* Cohort 2e: ROS1-positive solid tumor and progressed on any prior therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years (Cohort 2e only: Age ≥12 years).
2. Disease Criteria:

   1. Phase 1: Histologically or cytologically confirmed locally advanced or metastatic solid tumor with documented ROS1 rearrangement.
   2. Phase 2: Cohorts 2a, 2b, 2c and 2d: Histologically or cytologically confirmed locally advanced or metastatic NSCLC with ROS1 rearrangement.
   3. Phase 2: Cohort 2e: Histologically or cytologically confirmed locally advanced or metastatic solid tumor (other than NSCLC) with ROS1 rearrangement.
3. Prior anticancer treatment (except cohort 2a).
4. Phase 1: Must have evaluable disease (target or nontarget) according to RECIST 1.1. Phase 2: Must have measurable disease according to RECIST 1.1.
5. Adequate baseline organ function and bone marrow reserve.

Exclusion Criteria:

1. Patient's cancer has a known oncogenic driver alteration other than ROS1.
2. Known allergy/hypersensitivity to excipients of NVL-520.
3. Major surgery within 4 weeks of first dose of study drug.
4. Ongoing anticancer therapy.
5. Actively receiving systemic treatment or direct medical intervention on another therapeutic clinical study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 359 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) (Phase 1) | Within 28 days of last patient dosed during dose escalation
  Highest dose with dose-limiting toxicity (DLT) rate ≤ 25%
Recommended Phase 2 Dose (RP2D) | Within 28 days of last patient dosed during dose escalation.
  To determine the RP2D
Objective Response Rate (ORR) (Phase 2) | 2-3 years after first patient dosed.
  To determine ORR as assessed by BICR

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events, as assessed by CTCAE, v5.0 | Approximately 3 years.
  Incidence and severity of treatment-emergent adverse events (TEAEs)
Maximum plasma concentration (Cmax) of NVL-520 | Pre-dose and up to 24 hours post-dose
  To determine the maximum plasma concentration (Cmax) of NVL-520
Plasma concentration at the end of the dosing interval (Ctau) of NVL-520 | Pre-dose and up to 24 hours post-dose
  To determine the plasma concentration at the end of the dosing interval (Ctau) of NVL-520
Average plasma concentration (Cavg) of NVL-520 | Pre-dose and up to 24 hours post-dose
  To determine the average plasma concentration (Cavg) of NVL-520
Time of maximum concentration (Tmax) of NVL-520 | Pre-dose and up to 24 hours post-dose
  To determine the time of maximum concentration (Tmax) of NVL-520
Area under the curve at the end of the dosing interval (AUCtau) of NVL-520 | Pre-dose and up to 24 hours post-dose
  To determine the area under the curve at the end of the dosing interval (AUCtau) of NVL-520
Area under the curve from time 0 to 24 (AUC0-24) of NVL-520 | Pre-dose and up to 24 hours post-dose
  To determine the area under the curve from time 0 to 24 (AUC0-24) of NVL-520
Area under the curve from time 0 to infinity (AUCinf) of NVL-520 | Pre-dose and up to 24 hours post-dose
  To determine the area under the curve from time 0 to infinity (AUCinf) of NVL-520
Oral clearance (CL/F) of NVL-520 | Pre-dose and up to 24 hours post-dose
  To determine the oral clearance (CL/F) of NVL-520
Volume of distribution (Vz/F) of NVL-520 | Pre-dose and up to 24 hours post-dose
  To determine the volume of distribution (Vz/F) of NVL-520
Half-life (t1/2) of NVL-520 | Pre-dose and up to 24 hours post-dose
  To determine the half-life (t1/2) of NVL-520
Objective response rate (ORR) | 2-3 years after first patient dosed
  Determine ORR as assessed by BICR
Duration of response (DOR) | 2-3 years after first patient dosed
  Determine DOR of NVL-520 until radiographic disease progression or death
Clinical benefit rate (CBR) | 2-3 years after first patient dosed
  Determine CBR of NVL-520
Time to response | 2-3 years after first patient dosed
  Determine time to response of NVL-520
Progression-free survival (PFS) | Approximately 3 years
  Determine PFS of NVL-520 until radiographic disease progression or death
Overall survival (OS) | Approximately 3 years
  Determine OS
Rate of CNS progression | Approximately 3 years
  The incidence of CNS as first site of progression, alone or with concurrent extra-CNS progression
Intracranial objective response rate (IC-ORR) | Approximately 3 years
  Determine the intracranial objective response rate
Quality of life assessment using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | 2-3 years after first patient dosed
  EORTC QLQ-C30 measures cancer patients' physical, psychological, and social functions. Scale ranges from: 1, "Not at all"; 2, "A little"; 3, "Quite a bit"; to 4, "Very much." Higher score for the functioning scales and global health status denotes a better level of functioning, while higher scores on the symptom and single-item scales indicate a higher level of symptoms.
Quality of life assessment using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 29 module (EORTC QLQ-LC29) | 2-3 years after first patient dosed
  EORTC-QLQ-LC29 measures the quality of life in patients with lung cancer. Symptom scale ranges from: 1, "Not at all"; 2, "A little"; 3, "Quite a bit"; to 4, "Very much." For symptoms scales, higher scores indicated greater symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Upadhyay, MD, MBI, Study Director — Nuvalent Inc.
Locations (63):
- United States (20):
  - UCI Medical Center, Orange, California
  - Stanford Medicine, Palo Alto, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Miami, Coral Gables, Florida
  - University of Chicago, Chicago, Illinois
  - Mass General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - Ohio State University, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Washington / Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (2):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- University Hospital Leuven, Leuven, Belgium
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Research, Toronto, Ontario
- France (4):
  - Centre Legon Berard, Lyon
  - CHU de Nantes, Nantes
  - Claudius Regaud Institute, Toulouse
  - Institute Gustave Roussy, Villejuif
- Cologne University Hospital, Cologne, Germany
- Italy (7):
  - Università Politecnica Marche, Ancona
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - Istituto Europeo di Oncologia, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Oncologico Veneto, Padua
  - Ospedale Santa Maria delle Croci, Ravenna
  - Istituto Nazionale Tumori Regina Elena, Rome
- Japan (7):
  - Kanagawa Cancer Center, Kanagawa
  - Okayama University Hospital, Okayama
  - Kindai University Hospital, Osaka
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital Of JFCR, Tokyo
  - Wakayama Medical University Hospital, Wakayama
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - University Medical Centre Groningen, Groningen
- Singapore (2):
  - National University Hospital Singapore, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (4):
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - University Hospital of A Coruña, A Coruña
  - UOMI Cancer Center - Clinica Tres Torres, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - Gregorio Marañón Hospital, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
- Taiwan (3):
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (2):
  - Royal Marsden Hospital, London
  - Christie NHS Foundation Trust, Manchester